CLINICAL TRIAL: NCT04774237
Title: A 3-Dose, Multicenter, Randomized, Double-Masked, Crossover Phase 2 Safety and Efficacy Study of BRIMOCHOL™ Topical Ophthalmic Solution vs. BRIMOCHOL™ F Topical Ophthalmic Solution vs. Monotherapy With Carbachol Topical Ophthalmic Solution in Subjects With Emmetropic Phakic and Pseudophakic Presbyopia
Brief Title: Safety and Efficacy Study of BRIMOCHOL™, BRIMOCHOL™ F, and Carbachol in Subjects With Emmetropic Phakic and Pseudophakic Presbyopia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Visus Therapeutics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: VT-001
Record Dates: First submitted 2021-02-23; First posted 2021-03-01 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia | interventions — Carbachol; Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BRIMOCHOL™ (Experimental): A single drop in each eye at a visit.
  Interventions: Drug: BRIMOCHOL™
- BRIMOCHOL™ F (Experimental): A single drop in each eye at a visit.
  Interventions: Drug: BRIMOCHOL™ F
- Carbachol (Active Comparator): A single drop in each eye at a visit.
  Interventions: Drug: Carbachol

INTERVENTIONS:
Drug: BRIMOCHOL™ — A single drop in each eye at a visit.
  Other Names: carbachol/brimonidine tartrate
  Arms: BRIMOCHOL™
Drug: BRIMOCHOL™ F — A single drop in each eye at a visit.
  Other Names: carbachol/brimonidine tartrate
  Arms: BRIMOCHOL™ F
Drug: Carbachol — A single drop in each eye at a visit.
  Other Names: carbachol monotherapy
  Arms: Carbachol

SUMMARY:
Safety and Efficacy Study of BRIMOCHOL™ vs. BRIMOCHOL™ F vs. Carbachol Monotherapy Topical Ophthalmic Solutions in Subjects with Emmetropic Phakic and Pseudophakic Presbyopia

DETAILED DESCRIPTION:
A 3-Dose, Multicenter, Randomized, Double-Masked, Crossover Phase 2 Safety and Efficacy Study of BRIMOCHOL™ Topical Ophthalmic Solution vs. BRIMOCHOL™ F Topical Ophthalmic Solution vs. Monotherapy with Carbachol Topical Ophthalmic Solution in Subjects with Emmetropic Phakic and Pseudophakic Presbyopia

ELIGIBILITY:
Inclusion Criteria:

* Male or female in good general health
* Must have presbyopia

Exclusion Criteria:

* History of allergic reaction to the study drug or any of its components
* Any disease or medical condition that, in the opinion of the Investigator, would prevent the subject from participating in the study or might confound study results

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2021-10-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Global Research Management, Inc., Glendale, California
  - Eye Research Foundation, Newport Beach, California
  - Total Eye Care, PA, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- B, C, BF: Crossover design with 3 study treatments. Participants received Brimonidine, Carbachol PF, or BRIMOCHOL PF.
- B, BF, C: Crossover design with 3 study treatments. Participants received Brimonidine, BRIMOCHOL PF, or Carbachol PF.
- C, B, BF: Crossover design with 3 study treatments. Participants received Carbachol PF, Brimonidine, or BRIMOCHOL PF.
- C, BF, B: Crossover design with 3 study treatments. Participants received Carbachol PF, BRIMOCHOL PF, or Brimonidine
- BF, B, C: Crossover design with 3 study treatments. Participants received BRIMOCHOL PF, Brimonidine, or Carbachol PF.
- BF, C, B: Crossover design with 3 study treatments. Participants received BRIMOCHOL PF, Carbachol PF, or Brimonidine.
Period: Visit 2 First Intervention
Arm/Group | B, C, BF | B, BF, C | C, B, BF | C, BF, B | BF, B, C | BF, C, B
Started | 2 | 5 | 3 | 2 | 3 | 3
Completed | 2 | 5 | 3 | 2 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Period: First Washout
Arm/Group | B, C, BF | B, BF, C | C, B, BF | C, BF, B | BF, B, C | BF, C, B
Started | 2 | 5 | 3 | 2 | 2 | 3
Completed | 2 | 5 | 3 | 2 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Visit 3 Second Intervention
Arm/Group | B, C, BF | B, BF, C | C, B, BF | C, BF, B | BF, B, C | BF, C, B
Started | 2 | 5 | 3 | 2 | 2 | 3
Completed | 2 | 5 | 3 | 2 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Washout
Arm/Group | B, C, BF | B, BF, C | C, B, BF | C, BF, B | BF, B, C | BF, C, B
Started | 2 | 5 | 3 | 2 | 2 | 3
Completed | 2 | 5 | 3 | 2 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Visit 4 Third Intervention
Arm/Group | B, C, BF | B, BF, C | C, B, BF | C, BF, B | BF, B, C | BF, C, B
Started | 2 | 5 | 3 | 2 | 2 | 3
Completed | 2 | 5 | 3 | 2 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Single Drop Cohort: A single drop in each eye at a visit.
Arm/Group | Single Drop Cohort
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.3 (4.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 13
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With a >=15 Letter Gain Without a < 5 Letter Loss in Near Visual Acuity
Description: Primary Endpoint measured at Hour 1 post-dose at Study Visit - a Single drop Cohort
Time Frame: Day 1, Hour 1 post-dose
Measure: Count of Participants; unit: Participants
Groups:
- BRIMOCHOL; BRIMOCHOL PF; Carbachol PF: Single drop cohort
Arm/Group | BRIMOCHOL | BRIMOCHOL PF | Carbachol PF
Number analyzed (Participants) | 17 | 18 | 17
Participants | 15 | 15 | 16

2. Secondary Outcome: Change From Baseline ETDRS Letters Score in Distance Visual Acuity
Description: Secondary Endpoint measured at Hour 1 post-dose at Study Visit - a Single drop Cohort
Time Frame: Day 1, Hour 1 post-dose
Measure: Mean (Standard Deviation); unit: ETDRS letters
Groups:
- BRIMOCHOL™; BRIMOCHOL™ F; Carbachol: A single drop cohort
Arm/Group | BRIMOCHOL™ | BRIMOCHOL™ F | Carbachol
Number analyzed (Participants) | 17 | 18 | 17
ETDRS letters | 2.4 (3.39) | 2.8 (3.28) | 3.1 (2.86)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | BRIMOCHOL | BRIMOCHOL PF | Carbachol PF
All-Cause Mortality (participants affected / at risk) | 1/17 | 1/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 1/17 | 1/18 | 0/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BRIMOCHOL (N=17) | BRIMOCHOL PF (N=18) | Carbachol PF (N=17)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/37/NCT04774237/Prot_002.pdf
  • Statistical Analysis Plan (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT04774237/SAP_003.pdf